CLINICAL TRIAL: NCT07284602
Title: A Randomized, Double-Blind, Head-to-Head Phase 3 Trial to Evaluate the Efficacy and Safety of LYT-100 (Deupirfenidone) Compared to Pirfenidone at 52 Weeks in Adults With Idiopathic Pulmonary Fibrosis (SURPASS-IPF)
Brief Title: Trial to Evaluate the Efficacy and Safety of LYT-100 (Deupirfenidone) Compared to Pirfenidone in Adults With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: SURPASS-IPF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PureTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYT-100-2025-301; 2025-524493-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic Pulmonary Fibrosis; IPF; Pulmonary Fibrosis; Deupirfenidone; Pirfenidone; Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: Randomized double-blind treatment, 2 arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drugs are over-encapsulated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): deupirfenidone 825 mg TID
  Interventions: Drug: Deupirfenidone
- Active Comparator (Active Comparator): pirfenidone 801 mg TID
  Interventions: Drug: Pirfenidone (PFD)

INTERVENTIONS:
Drug: Deupirfenidone — size AA Swedish orange capsule
  Arms: Active
Drug: Pirfenidone (PFD) — size AA Swedish orange capsule
  Arms: Active Comparator

SUMMARY:
This is a study for adults with a lung disease called idiopathic pulmonary fibrosis. The main purpose of this study is to look at how well deupirfenidone improves lung function and how safe it is for people with idiopathic pulmonary fibrosis (IPF) when compared with pirfenidone. Participants may have been treated with an approved antifibrotic drug for up to a year in the past, but they cannot be on background antifibrotic treatment during this study. Participants will be randomly assigned (meaning by chance) to take either deupirfenidone or pirfenidone 3 times a day, and neither a participant nor their study team will know which study drug participants are on. Participants will be in the study for up to approximately 3 years. During the first year, participants visit the study site up to ten times and afterwards they visit the site every three months. All participants will remain on blinded study drug until the last participant has completed Week 52 Visit. They will have lung function tests, a check of their health, and will tell the study team about any unfavorable effects.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blind, head-to-head study comparing deupirfenidone 825 mg TID to pirfenidone 801 mg TID over 52 weeks of treatment in participants with IPF who are not on background therapy. This study is designed to demonstrate superior efficacy of deupirfenidone over pirfenidone as well as support the overall safety profile of deupirfenidone. Prospective participants will initially enter the Screening Period to determine study eligibility (Section 5). Eligible participants will be randomized 1:1 to receive either blinded deupirfenidone 825 mg TID or pirfenidone 801 mg TID as part of the Double-Blind Treatment Period for at least 52 weeks (Period 1). Depending on when participants enter the study, they may continue being treated for up to two more years (Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Is ≥40 years of age at the time of informed consent.
* Meets the diagnostic criteria of IPF American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Society (ALAT) 2022 guidelines.
* Has a maximum time from initial IPF diagnosis of 7 years.
* Has no prior exposure to pirfenidone or LYT-100, and has <12 months of prior exposure to nintedanib or any other approved antifibrotic therapies.
* Has definite or probable unusual interstitial pneumonia (UIP) on HRCT, performed within 12 months prior to Visit 1 and confirmed by the central reader.
* Has an FVC ≥45% of predicted normal at Visit 1.

Exclusion Criteria:

* Has, in the opinion of the Investigator, significant clinical worsening of IPF between Visit 1 and Visit 2.
* Has been hospitalized within 3 months prior to Visit 1 for acute exacerbation of IPF or other significant respiratory complication.
* Has prebronchodilator forced expiratory volume in 1 second (FEV1)/FVC <0.7 at Visit 1.
* Has a greater extent of emphysema vs fibrosis on the most recent HRCT scan as confirmed by the central reader.
* Has a diagnosis of any condition that could be an explanation for interstitial lung disease (ILD).
* Has a major extrapulmonary condition that could affect spirometry.
* Has a current diagnosis of other relevant respiratory disorders.
* Has significant pulmonary hypertension (PH).
* Has had a lung transplant.
* Has cardiovascular disease.
* Has underlying chronic liver disease/impairment.
* Has relevant chronic or acute infections including active viral hepatitis or poorly controlled HIV.
* Has had any major surgical procedures performed within 6 weeks prior to Visit 1 or is planning to have a major surgical procedure during the study.
* Has any documented active or suspected malignancy or history of malignancy within 5 years prior to Visit 1.
* Has any of the following laboratory abnormalities at Visit 1:

  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >1.5 × upper limit of normal (ULN).
  * Total bilirubin >1.5 × ULN. Exceptions may be made on a case-by-case basis for participants with Gilbert's syndrome in consultation with the Medical Monitor.
  * Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula.
* Is currently taking prednisone at a steady dose >10 mg/day or equivalent (a steady dose ≤10 mg/day is not exclusionary but the individual must be on a stable dose for at least 30 days prior to Visit 2).
* Use of any tobacco or combustible cannabis products within 3 months prior to Visit 1 or is unable to refrain from use during the trial.
* Has known symptoms of dysphagia, difficulty in swallowing capsules or tablets, or has had a total gastrectomy.
* Is currently enrolled in another clinical study (except observational/registry or biobank studies) or has used any investigational drug or device within 90 days prior to Visit 1.
* Has ever received stem cell therapy for the treatment of pulmonary fibrosis.
* Is currently pregnant, breastfeeding, or is planning to become pregnant during the study.
* Has had any prior exposure to LYT-100 or pirfenidone (even one dose).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Absolute change in forced vital capacity (FVC) measured in mL | Baseline to Week 52
  Evaluate the efficacy of deupirfenidone compared with pirfenidone on reduction in lung function decline in participants with IPF

SECONDARY OUTCOMES:
Absolute change in FVC percent predicted (FVCpp) | Baseline to Week 52
  Evaluate the efficacy of deupirfenidone compared with pirfenidone on reduction in lung function decline relative to individual predicted normal lung function

IPD SHARING:
Plan to Share IPD: No
Patient data protection laws in participating countries do not allow for IPD data sharing.